CLINICAL TRIAL: NCT00994019
Title: Short-term Natural History of Oral HPV Infection Among Young Adults
Brief Title: Study of Oral Papillomavirus In Teens and Twenties
Acronym: SPITT
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Principal Investigator, Gypsyamber D'Souza, Associate Professor, Johns Hopkins Bloomberg School of Public Health
Other Study IDs: 2422
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: STD
Keywords: HPV; oral cancer; young adults
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Recently human papillomavirus (HPV) has been recognized to cause some oropharyngeal (tonsil) cancer. But very little is known about oral HPV infection and risk factors. This study will evaluate how common oral HPV infection is, what sexual behaviors are associated with risk for infection, and how long infections tend to last.

DETAILED DESCRIPTION:
18-25 year old individuals are being recruited from STD clinics in Baltimore County and followed every three months for this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 -26 years

Exclusion Criteria:

* Never received HPV vaccine (Gardasil or Cervarix)

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: High risk young adults
Sampling Method: Non-Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2010-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Oral HPV infection | 24 months
  Oral rinse samples collected prospectively for 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Gypsyamber D'Souza, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- United States (2):
  - Baltimore County Woodlawn Health Centers, Baltimore, Maryland
  - Baltimore County Eastern Health Center, Baltimore, Maryland

REFERENCES:
- [Result] D'Souza G, Wentz A, Kluz N, Zhang Y, Sugar E, Youngfellow RM, Guo Y, Xiao W, Gillison ML. Sex Differences in Risk Factors and Natural History of Oral Human Papillomavirus Infection. J Infect Dis. 2016 Jun 15;213(12):1893-6. doi: 10.1093/infdis/jiw063. Epub 2016 Feb 10. PMID 26908748
- [Result] D'Souza G, Kluz N, Wentz A, Youngfellow RM, Griffioen A, Stammer E, Guo Y, Xiao W, Gillison ML. Oral Human Papillomavirus (HPV) Infection among Unvaccinated High-Risk Young Adults. Cancers (Basel). 2014 Aug 14;6(3):1691-704. doi: 10.3390/cancers6031691. PMID 25256827